CLINICAL TRIAL: NCT03855540
Title: AFISBIO - Atrial Fibrillation in Relationship to Sleep Quality and Plasma Biomarkers.
Brief Title: Atrial Fibrillation in Relationship to Sleep Quality and Plasma Biomarkers
Acronym: AFISBIO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Premedix Academy (Other)
Responsible Party: Sponsor
Other Study IDs: 0012018
Record Dates: First submitted 2018-12-05; First posted 2019-02-26 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; ECG monitoring; quality of sleep; plasmatic biomarkers
MeSH Terms: conditions — Atrial Fibrillation; Sleep Initiation and Maintenance Disorders | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Adult patients with documented paroxysmal, nonvalvular atrial fibrillation with CHA2DS2-VASc score > 2 (for females > 3) and sinus rhythm at the time of inclusion. In total 100 patients will be included.
  Interventions: Diagnostic Test: ECHOcardiography; Diagnostic Test: Peripheral blood samples for plasmatic biomarkers; Diagnostic Test: Athens insomnia scale questionnaire
- Control group: Patients without a history of palpitations or irregular heart rhythm. AFib will be excluded with the help of 7 days ECG Holter and ECG event recorder monitoring. In total 100 patients will be included.
  Propensity matching according to the:
  * CHA2DS2-VASc parameters
  * LVEF: preserved (<40%), mid-range (40-49%) and reduced (>50%)
  * Presence of diastolic dysfunction
  * Glomerular filtration rate: (≥1,5 ml/s), (1,4-1 ml/s) and (0,9-0,5 ml/s)
  * Drugs: ACE-I/ARB, betablockers, digoxin, amiodarone
  * BMI: (<30kg/m2), (30-39kg/m2) and (≥40kg/m2)
  * Smoking (>5 cigarettes per day)
  Interventions: Diagnostic Test: ECHOcardiography; Diagnostic Test: Peripheral blood samples for plasmatic biomarkers; Diagnostic Test: Athens insomnia scale questionnaire; Diagnostic Test: ECG Holter monitor; Diagnostic Test: ECG event recorder

INTERVENTIONS:
Diagnostic Test: ECHOcardiography — ECHO parameters
  1. LA diameter
  2. LVEDD
  3. LVEF
  4. Diastolic dysfunction
  5. Valvular disease
Diagnostic Test: Peripheral blood samples for plasmatic biomarkers — 1. Coagulation
     * D - dimer
     * Fibrinogen
  2. Inflammation and fibrosis
     * Hs - CRP
     * AGEs
     * Soluble RAGE
  3. Hemodynamics (LA stretch)
     * Apelin
     * NT - proBNP
     * Hs - troponin
  4. MiRNA
     * miRNA - 1
     * miRNA - 133
     * miRNA - 29b
     * miRNA - 208a
     * miRNA - 208b
     * miRNA - 499
Diagnostic Test: Athens insomnia scale questionnaire — Athens insomnia scale questionnaire
Diagnostic Test: ECG Holter monitor — Patient receives ECG Holter monitor if included to the control group
  Groups: Control group
Diagnostic Test: ECG event recorder — Patient receives ECG event recorder for twice daily (or if symptoms), 90 seconds duration ECG monitoring if included to the control group
  Groups: Control group

SUMMARY:
A. Compare the plasmatic biomarkers between the cohort with and without AFib.

B. Find sensitive and specific biomarkers that could be used for the diagnostic management of AFib.

C. Compare the quality of sleep between the cohort with and without AFib by the means of sleeping quality questionnaire

DETAILED DESCRIPTION:
AFib is the most common sustained arrhythmia, associated with an increased risk of stroke, heart failure, and mortality. Despite the high prevalence, AFib may be asymptomatic and consequently subclinical. Detection of subclinical AFib is highly challenging as only a minority of the patients is diagnosed during a standard examinations with a 12 - lead ECG or a 24h ECG Holter monitoring. Documented AFib causes 15% of ischemic strokes, however approximately 25% of ischemic strokes is of an unknown etiology. It is believed that undetected subclinical AFib is responsible for these strokes. There is also evidence that asymptomatic AFib is associated with a higher incidence of strokes in comparison to symptomatic AFib.

Due to the fact that the standard ECG examination is not sufficient for AFib detection, various ECG screening methods have been introduced. Intermittent short ECG recording seems to be more effective than 24-hour Holter ECG in the detection of the arrhythmia however, it is not known whether it is superior to the 7 - day ECG Holter monitoring.

Plasmatic biomarkers might be of a paramount importance in the diagnostic management.

Several plasmatic biomarkers were tested to find an association with AFib. Perhaps the most studied ones were the natriuretic peptides that showed to be significantly increased in patients with AFib. Similarly, high sensitivity troponins are elevated in patients with the AFib. Another marker of left atrial stretching and also of ionotropic effects is apelin. Patients with lone AFib showed a significantly decreased levels of this peptide. Conflicting results were shown in studies with inflammatory biomarkers such as high sensitivity CRP Parameters reflecting thrombogenesis were also found to be associated with the arrhythmia. Fibrinogen and fibrin D-dimer were significantly increased in paroxysmal AFib. Finally, in the last years, the circulating micro RNAs emerged as a promising biomarker of AFib, having important function in suppression of messenger RNA responsible for thrombogenesis and ionotropic functions.

The weakness of the mentioned studies is, that the biomarkers were usually tested in patients with a few comorbidities. So, it is not known whether these biomarkers are specific for AFib "per se" or whether they just reflect pathophysiological mechanisms like inflammation, fibrogenesis or left atrium stretching that is also present in other cardiovascular diseases. Furthermore, the AFib cohorts were often not matched with the control groups adding more uncertainty. To clarify these questions, we designed a study where plasmatic biomarkers will be studied in high risk cohort of patients with AFib having several cardiovascular comorbidities. These patients will be subsequently matched with a control group according to the age, gender and the cardiovascular comorbidities.

Similarly, as the continuum of organic changes of the heart from the left ventricular diastolic dysfunction, left atrial dilatation ending with heart failure, there is also "arrhythmology continuum" in patients with arterial hypertension to supraventricular premature contractions via paroxysmal tachycardia of fibrillation up to the permanent atrial fibrillation (AFib). A common etiopathology factor of these disorders is increased sympathetic activity, which together with the catecholamine release during the stress causes arrhythmogenic substrates due to the atrial fibrogenesis. The relation between sleep disorders and the AFib is poorly understood. Micro awakenings during the night increases sympathetic activity and the arterial blood pressure. Other possible mechanism might be the decrease of plasmatic melatonin related to aging. Sleep disorders are linked to the increased heart rate, worsening of the heart rate variability, increased metabolism and body temperature, increased beta EEG activity and activation of the hypothalamic - pituitary - adrenal axis. In patients with arterial hypertension, there is an increased occurrence of premature atrial contractions that is linked to increased risk of AF incidence.

ELIGIBILITY:
Inclusion Criteria: The specific criteria for inclusion in the study group are:

* Age >17 years
* Documented, nonvalvular paroxysmal AFib in the duration of more than 6 min. (medical history or ECG monitoring)
* CHA2DS2-VASc score > 2 for males
* CHA2DS2-VASc score > 3 for females
* Sinus rhythm at the time of inclusion

The specific criteria for inclusion in the control group are:

* No history of palpitations
* AFib exclusion with the 7 days ECG Holter and ECG event recorder monitoring
* Propensity matching

Exclusion Criteria: Exclusion criteria for both groups:

* Electrical cardioversion less than 7 days prior to inclusion
* Acute coronary syndrome less than 1 month prior to inclusion
* Cardiac surgery less than 3 months prior to inclusion
* Acute or decompensated heart failureat the time of inclusion
* Pregnancy
* Cardiomyopathy
* Alcoholism (≥ 8 drinks/week)
* Thyrotoxicosis
* Renal Disease (Dialysis/ transplant/CrCl < 0,5ml/s)
* Liver disease (cirrhosis/ transaminase > 3x ULT/ bilirubin > 2x ULT)
* Mechanical proshetic valves
* Severe mitral stenosis
* Class I and IV antiarrhythmic drugs usage in last month
* Class III antiarrhythmic drugs usagein last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Slovak hospitals and outpatients clinics
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-04-11 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Plasmatic biomarkers | Day of inclusion
  Compare the plasmatic biomarkers between the cohort with and without atrial fibrillation:
  1. Coagulation a D - dimer b Fibrinogen
  2. Inflammation and fibrosis a Hs - CRP b AGEs c Soluble RAGE
  3. Hemodynamics (LA stretch) a Apelin b NT - proBNP c Hs - troponin
  4. MicroRNA a miRNA - 1 b miRNA - 19 c miRNA - 21 d miRNA - 124 e miRNA - 150 f miRNA - 328
Quality of sleep | Day of inclusion
  Compare the quality of sleep between the cohort with and without atrial fibrillation by the means of Athens Insomnia Scale (AIS). It is measured by assessing eight factors amongst which first five factors are related to nocturnal sleep and last three factors are related to daytime dysfunction. These are rated on a 0-3 scale and the sleep is finally evaluated from the cumulative score of all factors and reported as an individual's sleep outcome. A cut-off score of ≥6 on the AIS is used to establish the diagnosis of insomnia.

SECONDARY OUTCOMES:
Diagnostic plasmatic biomarker | Day of inclusion
  Find sensitive and specific biomarker that could be used for the diagnostic management of atrial fibrillation:
  1. Coagulation a D - dimer b Fibrinogen
  2. Inflammation and fibrosis a Hs - CRP b AGEs c Soluble RAGE
  3. Hemodynamics (LA stretch) a Apelin b NT - proBNP c Hs - troponin
  4. MicroRNA a miRNA - 1 b miRNA - 19 c miRNA - 21 d miRNA - 124 e miRNA - 150 f miRNA - 328

CONTACTS AND LOCATIONS:
Overall Officials: Allan Bohm, MD, Principal Investigator — The National Institution of Cardiovascular Diseases; Stefan Farsky, Associate professor, Principal Investigator — Slovak league against hypertension
Locations (4):
- Slovakia (4):
  - Allan Bohm, Bratislava
  - East Slovak Institute of Cardiovascular Diseases, Košice
  - Hospital, Malacky
  - University hospital, Nitra

IPD SHARING:
Plan to Share IPD: No